CLINICAL TRIAL: NCT04525989
Title: Preoperative Short-Course Radiation Therapy With PROtons Compared to Photons In High-Risk RECTal Cancer (PRORECT): A Prospective Randomized Swedish Phase II Trial
Brief Title: Preoperative Short-Course Radiation Therapy With PROtons Compared to Photons In High-Risk RECTal Cancer (PRORECT)
Acronym: PRORECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Valdman (Other)
Responsible Party: Sponsor-Investigator, Alexander Valdman, MD, PhD, Senior Consultant Radiation Oncologist, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRORECT
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Proton therapy; Preoperative radiation; Short-course; Primary adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proton therapy (Experimental): 5 x 5 Gy External radiation therapy with Protons
  Interventions: Radiation: Radiation therapy
- Photon therapy (Active Comparator): 5 x 5 Gy External radiation therapy with Photons
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — 5 x 5 Gy external radiation therapy

SUMMARY:
To investigate a potential toxicity benefit of preoperative radiation therapy with protons compared to conventional photon beam radiation therapy in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether proton beam radiotherapy in locally advanced rectal cancer can offer meaningful reductions in acute gastrointestinal toxicity compared to standard treatment with photons which may improve patient's tolerability of neoadjuvant chemotherapy.

There are currently no published clinical reports evaluating the use of proton therapy in the upfront treatment of locally advanced rectal cancer. There are further no published randomized trials comparing radiotherapy with photon vs proton in locally advanced rectal cancer.

This is a prospective randomized trial, initially run at the limited number of centres but later expanded to other centres participating in the Skandion network. Patients will be treated with short course 5 x 5 Gy radiation scheme with either photons (standard arm) or protons (Skandion clinic) followed by four to six cycles of combination chemotherapy (capecitabine and oxaliplatin) and surgery. The rectal tumour will be removed by TME/PME surgery or more extensive surgery if required because of tumour extent.

All patients will receive at least 4 courses of CAPOX (Capecitabine b.i.d.1000 mg/m2 day 1-14 every 3 weeks, Oxaliplatin 130 mg/m2 day 1 every 3 weeks) week 3-14, followed by surgery at week 17-20.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Primary tumour characteristics

* Biopsy-proven, newly diagnosed primary rectal adenocarcinoma, i.e. with the lowest part of the tumour less than 16 cm from the anal verge detected using a rigid rectoscope.
* Locally advanced tumour fulfilling at least one of the following criteria on pelvic MRI indicating high risk of failing locally and/or systemically:

  * Clinical stage (c) T4b, i.e. infiltration of an adjacent organ or structure like the prostate, urinary bladder, uterus, sacrum, pelvic floor or side-wall (according to TNM version 8).
  * cT4a, i.e. peritoneal involvement.
  * Extramural vascular invasion (EMVI+).
  * N2-status regarded as metastatic according to ESGAR consensus criteria
  * Positive MRF, i.e. tumor or lymph node one mm or less from the mesorectal fascia.
  * Metastatic lateral nodes (lat LN+) according to ESGAR consensus criteria

Inclusion Criteria - General

* Staging done within 6 weeks before start of radiotherapy. No contraindications to chemotherapy with CAPOX including adequate blood counts, (within 5 weeks prior to randomisation):

  * white blood count ≥4.0 x 10*9/L
  * platelet count ≥100 x 10*9/L
  * clinically acceptable haemoglobin levels
  * creatinine levels indicating renal clearance of ≥50 ml/min
  * bilirubin ˂35 µmol/l.
* ECOG performance score ≤1
* Patient is considered to be mentally and physically fit for chemotherapy with CAPOX as judged by the oncologist.
* Age ≥18 years
* Written informed consent.
* Adequate potential for follow-up.

Exclusion Criteria:

* Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen.
* Presence of metastatic disease or recurrent rectal tumour. Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis.
* Concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years.
* Known DPD deficiency.
* Any contraindications to MRI (e.g. patients with pacemakers).
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Concurrent uncontrolled medical conditions.
* Any investigational treatment for rectal cancer within the past month.
* Pregnancy or breast feeding.
* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia, e.g. atrial fibrillation, even if controlled with medication) or myocardial infarction within the past 12 months.
* Patients with symptoms of peripheral neuropathy.
* Patients with pacemaker or ICD
* Patients with bilateral hip protheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute grade 2-5 gastrointestinal toxicity | From start of radiotherapy to planned start of the third (3) CAPOX cycle (week 9-10 of the trial)
  The incidence of acute preoperative grade 2-5 gastrointestinal toxicity according to CTCAE v5.0 associated with proton vs. photon radiotherapy

SECONDARY OUTCOMES:
Incidence of grade >2 hematologic and non-hematologic toxicity | Baseline up to five years after treatment
  The incidence of grade >2 hematologic (blood count, febrile neutropenia) and non-hematologic toxicity (general, genitourinary, gastrointestinal, skin) associated with protocol treatment, assessed by CTCAE v5.0 in the preoperative period, the postoperative period, and overall.
  Patient reported side-effects will be assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire, the QLQ-C30, version 3. The QLQ-C30 will be supplemented with the disease specific module (rectal-cancer) QLQ-CR29. During radiotherapy, daily reported symptoms will be investigated by a newly developed symptom scale, Radiotherapy related symptom assessment scale (RSAS). The questionnaire includes 13 items specific for current diagnose. The RSAS is a validated instrument for assessing symptom intensity and distress in patients with different cancer disease undergoing radiotherapy, with psychometric properties within the expected range.
Differences in patient reported outcomes (PRO) | Baseline, Day 1-5, 2 and 3 weeks, 3, 6, 9, 12, 24, 36 and 60 months
  Differences in patient reported outcomes (PRO) between treatment arms in the preoperative period, the postoperative period, and overall
Proportion of patients being able to undergo full dose neoadjuvant chemotherapy | From week 3 until week 20 of the trial
  Differences between treatment arms in proportion of patients being able to undergo full dose neoadjuvant chemotherapy i.e. at least 4 cycles of CAPOX or 6 cycles of FOLFOX
Tumour regression grading (mrTRG) | Baseline to response evaluation week 16-17 of the trial
  Radiological assessment and comparison of tumour regression grading (mrTRG) between treatment arms
Cost effectiveness analysis measured by QALY | Time from randomization up to 5 years
  Health economic comparison between proton and photon treatment. Cost effectiveness analysis measured by QALY

OTHER OUTCOMES:
Disease free survival | Time from randomization until first recurrence, local/regional/systemic or death
  Disease free survival after proton vs. photon treatment
Overall survival | Time from randomization until death
  Overall survival after proton vs. photon treatment
Quality of Life (QLQ-C30) | Baseline, 3 weeks, 3, 6, 9, 12, 24, 36 and 60 months
  Quality of life after proton vs. photon treatment (QLQ-C30)
Difference in postoperative complications | From week 17-20 of the trial up to 5 years
  Difference in postoperative complications between study arms measured by LARS score
Clinical complete remission (cCR) | From start of treatment up to 1 year
  Proportion of patients who reach a clinical complete remission (cCR), enter a watch-and-wait period and remain free of regrowth at least one year
Incidence of acute lumbar plexus neuralgia | From baseline until week 4 of the trial
  Difference between treatment arms in acute lumbar plexus neuralgia grade 1-3 measured as a change from baseline according to CTCAE 5.0
Exploratory: Concentrations of CD8+ and FOXP3 + tumour-infiltrating T cells | Postoperative pathology from week 17 until week 24 of the trial
  Difference between treatment arms in concentrations of CD8+ and FOXP3 + tumour-infiltrating T cells after given radiotherapy
Exploratory: Difference in concentrations of CEA (carcinoembryonic antigen) between treatment arms | CEA measurements at baseline, week 3, 6, 9 and 12 of the trial
  Change from baseline in concentrations of circulating CEA (carcinoembryonic antigen) between treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Valdman, MD, PhD, Principal Investigator — Department of Radiotherapy, Karolinska University Hospital, Stockholm, Sweden
Locations (9):
- Sweden (9):
  - Karolinska University Hospital, Theme Cancer, Dept of Pelvic cancer, Stockholm, Solna
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Stockholm South General Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedone C, Sorcini B, Staff C, Farlin J, Fokstuen T, Frodin JE, Nilsson PJ, Martling A, Valdman A. Preoperative short-course radiation therapy with PROtons compared to photons in high-risk RECTal cancer (PRORECT): Initial dosimetric experience. Clin Transl Radiat Oncol. 2022 Dec 17;39:100562. doi: 10.1016/j.ctro.2022.100562. eCollection 2023 Mar. PMID 36582423